CLINICAL TRIAL: NCT05706571
Title: The Effect of Augmented Reality and Benner Model-Based Teaching on Nursing Students' Learning: Child Patient End-of-Life Care Module
Brief Title: Child Patient End-of-Life Care Module
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Makbule Yılmaz, nurse, Medipol University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: MedipolU-makbule-yılmaz-001
Record Dates: First submitted 2023-01-23; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Pediatric Asthma
Keywords: terminal care; nursing; Benner
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Nicel ve nitel verilerin oluşturulmasında ikisi deney ve biri kontrol grubu olmak üzere üç grupta oluşacaktır. Araştırmanın deney ve kontrol grupları oluşturulurken seçkisiz, yansız seçim yapılarak gruplar arasında homojenlik sağlanması planlanmaktadır. Arttırılmış gerçeklik ve Benner modeli ile öğretimin hemşirelik öğrencilerinin çocuk hasta yaşam sonu bakım modülünü deney ve kontrol gruplarına herhangi bir uygulama yapmadan önce ön test yapılması planlanmaktadır. Son testler ise kontrol grubuna; klasik öğrenme, deney 1 grubuna; Benner'n Acemilikte Uzmanlığa Modeline göre simülasyon sonrası, deney2 grubuna ise mobil arttırılmış gerçeklik uygulaması sonrası son testlerin yapılması planlanmaktadır.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control grup (skill laboratory) (No Intervention): The control group of the study: The control group of the study; Students will be formed from students whose school number has a single last digit. The experimental 1 group and control group of experimental 2 groups of the study consist of the same group. Before the theoretical lecture of the pediatric patient end-of-life care module of nursing students teaching with augmented reality and the Benner model, students will be pre-tested. After the pre-test, students are taught on a virtual case in the last hours and days of life; Theoretical lecture will be given by the researcher in the form of a PowerPoint presentation, which will last 60 minutes, using question-answer, discussion, and commentary methods. A final test will be given at the end of the course.
- experimental group1 (Benner model) (Experimental): Experiment 1 Group of the Research With the Benner model, it is planned to create the pediatric end-of-life care module for nursing students in the Fall Term of the 2023-2024 Academic Year, with an estimated 140 students enrolled in the Istanbul Medipol University Faculty of Health Sciences Nursing Department Child Health and Diseases Nursing Course. The enrolled students will form the novice nurse group according to the Benner model of the research. A pre-test will be done before the theoretical lesson is given to the novice nurse group of the research.
  Interventions: Other: control group (skill laboratory), experimental group 1 (Banner model) and experimental group2 (augmented reality mobile application)
- experimental group2 (augmented reality mobile application) (Experimental): Application of the Research to the Experimental Group 2 Experiment 2 group of the research; In the Fall Term of the 2023-2024 Academic Year, an estimated 140 students will be enrolled in the Istanbul Medipol University Health Sciences Faculty Nursing Department Child Health and Diseases Nursing Course. The 3rd group of the study will be pre-tested before the theoretical lecture of the Pediatric Patient End-of-Life Care Module with the augmented reality method and Benner model. At the end of the pre-test, students will be given a theoretical lecture.
  Interventions: Other: control group (skill laboratory), experimental group 1 (Banner model) and experimental group2 (augmented reality mobile application)

INTERVENTIONS:
Other: control group (skill laboratory), experimental group 1 (Banner model) and experimental group2 (augmented reality mobile application) — In the research, the control group will form the control group of both experiment one and experiment two. In the creation of quantitative and qualitative data, it will be formed in three groups, two of which are the experimental group and one is the control group. While forming the experimental and control groups of the research, it is planned to ensure homogeneity between the groups by making random and unbiased selection. It is planned to do a pre-test before applying the child patient end-of-life care module of nursing students of teaching with augmented reality and Benner model to the experimental and control groups.
  Arms: experimental group1 (Benner model); experimental group2 (augmented reality mobile application)

SUMMARY:
This research is planned to be carried out by using a mixed method that combines quantitative and qualitative approaches to investigate the effect of teaching with augmented reality and the Benner model on the learning of the pediatric end-of-life care module of nursing students.

The population of the research will be approximately 140 students who are enrolled in Istanbul Medipol University Faculty of Health Sciences Nursing Department Child Health and Diseases Nursing Course in the Fall Term of the 2023-2024 Academic Year. Since it is aimed to reach the universe in the study, sample selection will not be made.

Data collection tools of the research; "Descriptive Characteristics Form", "Pediatric Patient End of Life Care Module Knowledge Test", and "Tanatophobia Scale" will be administered to the control and experimental groups before and after the application. "Child Patient End of Life Care Module Evaluation Guide" and "Semi-Structured Interview Form" will be given to the experimental groups after the application, while the "Augmented Reality Evaluation Form" and the E-Learning Attitude Scale are planned to be administered only to the experimental2 group. A quasi-experimental design with the pretest-posttest control group, one of the quantitative research methods, will be applied. Qualitative data, on the other hand, will be administered to the experimental groups in the form of a focus group interview with a "Semi-Structured Interview Form". In the research, the control group will form the control group of both experiment one and experiment two.

After the research, teaching the Child Patient End-of-Life Care module according to Augmented Reality and Benner model, increasing the professional skill performance/academic success level of the students who improve the knowledge and skill levels of the nurse students before they go to the clinical area, orienting the student to learn by experimenting with three-dimensional visual/auditory animations, In a complicated end-of-life situation, it is aimed to increase the stress, motivation and skill competence of the student before the clinical environment to the "expert level at the beginner level", with fast decision making and a realistic education environment.

DETAILED DESCRIPTION:
Introduction Description of the Subject/ Problem Status The end-of-life period is the period in which health declines due to the last stage of the disease, the organism loses its ability to renew itself, and the state of being alive ends. This process affects both the family and the patient in many ways. Meeting the physical, spiritual, psychological, and cultural needs of the family and the patient in the last days and hours of life reflects the nurse's holistic care.

The first step towards becoming a skilled clinician and advocacy guide for the nurse who cares for the sick individual in the last days and hours of life is to have a clear understanding of what care the patient and family want at the end of life . The basic desires of patients and families at the end of life. It is process-oriented and relationship-based rather than focusing on medical goals. In addition, patients prefer to die at home (Tang, 2003), symptom management and communication management of a specialist healthcare professional in reporting bad news are among the important themes of end-of-life care.

To provide evidence-based care in nursing education, expert educators use patients created with simulation-based virtual reality methods, high-quality human simulators, standardized patients, augmented reality, and virtually created patients . Virtual reality can artificially recreate all senses, and experiences, including sight, hearing, touch, and smell. Augmented reality tries to replace reality by bridging "virtual and real worlds" (Wu H-K, Lee SW-Y, Chang H-Y, Liang J-C. 2013; Ferguson, C., Davidson, P. M., Scott, P. J., Jackson, D., &Hickman, L. D. (2015) These methods help students provide appropriate nursing care safely and efficiently without fear of their professional skills and knowledge.

The use of simulation in nursing education is an integral part of the curriculum and will demonstrate the benefit of learning to nurse students of all levels. The next phase of simulation-based learning is the wide variety of new technologies currently available, including virtual and augmented reality. The use of these new technologies will bring the need for standard definitions, assessment of the impact on learning, and new opportunities for research. By incorporating virtual and augmented reality into the curricula of nurse academicians, simulation-based learning methods will provide an opportunity to create a new era in education.

While providing care for the individual in the last days and hours of life, it is very difficult for nurses to control the individual's own feelings about the death process when the individual suffers, and works with families in an extremely difficult time . Nurses' training on pediatric end-of-life care includes a wide variety of modules, including didactic sessions, supervised clinical practice, mentoring, role-playing of predetermined scenarios, simulated/standardized patient encounters, computer-based gaming, augmented reality (AR), and virtual reality (VR) modules. teaching methods are used . Academics and nurses have to adjust the experiences they learn in many different ways to suit the student. Augmented reality (AR), virtual reality (SG), and play all provide an immersive student experience where new ways of learning are needed more than ever before. will be used in many settings to optimize care and improve the health outcomes of individuals in all care settings.

A theoretical foundation will be needed if the simulation is to continue to progress as a discipline. Benner's "Novice to Expert Model" will provide the necessary conceptual structure to guide simulation facilitator development and aid understanding of the learning path. Although individuals who use the simulation are experts in their clinical fields, they go back to the novice stage when they start to practice. This model-based approach, which defines and implements the developmental stage of nurses (Novice, Competence, Competence, Mastery, and Expertise), will serve as a guide for simulation education-training programs and infrastructure Purpose of the study This study will be carried out to determine the effect of teaching with augmented reality and the Benner model on the learning of the pediatric end-of-life care module of nursing students.

Study Hypotheses/goals H0 -1: Teaching the Pediatric Patient End of Life Care module with Augmented Reality Method has no effect on the student's level of knowledge.

H1-1: Teaching the Child Patient End of Life Care module with Augmented Reality Method affects the student's level of knowledge.

H0 -2: Teaching the Pediatric Patient End of Life Care module with Augmented Reality Method does not affect the student's practice skill time.

H1-2: Teaching the Pediatric Patient End of Life Care module with Augmented Reality Method affects the student's practice skill time.

H0 -3: Teaching the Pediatric Patient End of Life Care module with the Benner Model has no effect on the student's level of knowledge.

H1-3: Teaching the Pediatric Patient End of Life Care module with the Benner Model affects the student's level of knowledge.

H0 -4: Teaching the Pediatric Patient End of Life Care module with the Benner Model does not affect the student's practice skill level.

H1-4: Teaching the Pediatric Patient End of Life Care module with the Benner Model affects the student's practice skill level.

H0 -5: Teaching the Pediatric Patient End-of-Life Care module with the direct instruction method does not affect the student's level of knowledge.

H1-5: Teaching the Pediatric Patient End-of-Life Care module with the direct instruction method affects the student's level of knowledge.

Importance of the Study The complex nature of pediatric end-of-life care requires extensive training for nurses working with children and their families in life-threatening conditions. Knowledge of evidence-based best practices is an essential component of this training. However, due to the nature of working with a vulnerable population, additional educational elements will be required for quality care .

Simulation-based learning on virtual patients is a widely accepted teaching method in nursing education. It bridges theory and practice and provides the opportunity for novice nursing students to practice the skills necessary for practice in a safe environment. Novice students do not have the experience or context to form the clear mental picture or image required for simulated scenarios. (Vaughn, J., Lister, M., & Shaw, RJ (2016). Mobile applications such as AG/SG in simulated patients will give novice clinicians a chance to subvert a group of virtual patients before taking on a live patient.This study will provide novice nurses with a roadmap on how to approach patients with AR application.

Among the evidence-based practices in nursing education, another education will provide theory and model-based care to the individual. Benner's "Novice to Expert Model" provides the necessary conceptual structure to guide the facilitator's development of simulation and aid understanding of the learning path. In Benner's model, experience, education, and clinical knowledge development were discussed in determining the competency levels of nurses. End-of-life care modules provide holistic care for the needs of the child and family. These modules include evidence-based practice, family-centered care, The cultural values of the patient and family, the grieving process, symptom management, and communication methods in reporting bad news will be a guide in the study.

Many educational technologies that change the social structure in the twenty-first century are constantly being renewed and developed. As new educational technologies develop, different learning methods from classical learning methods develop. One of these methods is the augmented reality method. Augmented reality application provides theoretical and practical training as a whole in nursing education to prepare the student for professional life in end-of-life care and to give the student a professional nursing identity. In this study; With the augmented reality application, it is expected that the student's affective, cognitive and psychomotor skills will be improved. Students will be able to use these skills wherever they want with the application installed on their mobile phones without entering the laboratory environment. Depending on the learning in end-of-life care based on the Benner model with augmented reality method, the student; when he/she starts clinical practice, he/she will be provided to develop clinical wisdom and clinical decision-making skills. In addition, the augmented reality application, increases the professional skill performance / academic success level of the students, directing the student to learn by experimenting with three-dimensional audio / visual animations, quick decision-making in a complicated end-of-life situation, and a realistic educational environment. it is aimed to increase the skill competence to the level of "expertise at the novice level".

Material and method of the research:

Purpose and Type of Research This research is planned to be conducted in a mixed-method study in which quantitative and qualitative approaches are included in order to investigate the effect of teaching with augmented reality and the Benner model on the learning of the pediatric end-of-life care module of nursing students.

Place and Time of Research The research is planned to be carried out within the scope of the Istanbul Medipol University Faculty of Health Sciences Child Health and Diseases Nursing practice course in the Fall Term of the 2022-2023 and 2023-2024 Academic Years.

ELIGIBILITY:
Inclusion Criteria:

* • Must have taken the course in child health and diseases nursing,

  * Child health and diseases nursing language students
  * Voluntary participation in the study,
  * Internet access,
  * The phones on which the augmented virtual reality application will be installed must be Android,
  * Not having lost a first-degree relative recently,

Exclusion Criteria:

Reasons for being excluded from the study:

* Not participating in demonstrations and group practices
* Health vocational high school students
* Not attending the lecture
* Not participating in augmented virtual reality application

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Child Patient End of Life Care Module Knowledge Test | one week
  In order to prepare the Pediatric Patient End-of-Life Care Module Knowledge Test, the theoretical course content of the Pediatric End-of-Life Care Module was created by the researcher in accordance with the literature on Benner's Novice to Expertise Model and end-of-life care in the last days and hours of life.
Thanatophobia Scale | one week
  Çiftçioğlu and Seren (2019) Turkish validity and reliability of the Thanatophobia (Fear of Death) scale was created by Merrill et al. The Thanatophobia scale has a total of 7 items. The items of the scale are likert type, starting from 1 to 7 in the "strongly disagree" category and scored towards the "strongly agree" category. The individual's score on the scale is directly proportional to the fear of death.

SECONDARY OUTCOMES:
Attitude Scale Towards E-Learning | one month
  The scale developed by Haznedar and Baran in order to determine students' attitudes towards e-learning in higher education institutions consists of 20 items. The sub-dimensions of the scale; 10 items of "Susceptibility to E-Learning" (1,5,6,7,9,12,15,16,17,20) and 10 other items of "E-Learning Avoidance" (2,3,4,8,10, 11,13,14).
Augmented Reality Applications Attitude Scale | one month
  Small et al. (2014) "Augmented Reality Applications Attitude Scale" consists of 15 items. 15 items in the scale; 7 items (1, 4, 5, 7, 9, 11, and 15) included the Satisfaction with Use sub-factor, 6 items (2, 3, 6, 8, 10, and 14) the Use Anxiety sub-factor, and 2 items (12 and 13). It measures the Willingness to Use sub-factor. The scale consists of a 5-point Likert structure.
Augmented Reality Evaluation Form | one month
  "Augmented Reality Evaluation Form" was prepared by the researcher in accordance with the literature.
Structured Interview form | one month
  A focus group interview is a qualitative data collection method, which is generally held with 4-12 participants and a moderator and aims to collect data by creating a polyphonic environment where participants do not need to hide their true thoughts.

CONTACTS AND LOCATIONS:
Overall Officials: Sema Kuguoğlu, Prof.Dr., Study Chair — Medipol Unıversty

IPD SHARING:
Plan to Share IPD: No